CLINICAL TRIAL: NCT00655642
Title: A Randomized, Double Blind, and Placebo-Controlled Trial Comparing Ondansetron, Metoclopramide and Promethazine for the Treatment of Nausea and Vomiting in the Adult Emergency Department.
Brief Title: Comparison of Ondansetron, Metoclopramide and Promethazine for the Treatment of Nausea and Vomiting in the Adult ED
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Conditional analysis showed observed differences were significantly less than power calculations
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Tyler Barrett, Assistant Professor of Emergency Medicine, Vanderbilt University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VUMC 0612369
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Results first posted 2011-05-09 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-09

CONDITIONS: Nausea
MeSH Terms: conditions — Nausea | interventions — Ondansetron; Metoclopramide; Promethazine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Ondansetron (Active Comparator): Ondansetron 4 mg intravenous administration
  Interventions: Drug: Ondansetron
- Metoclopramide (Active Comparator): Metoclopramide 10 mg intravenous administration
  Interventions: Drug: Metoclopramide
- Promethazine (Active Comparator): Promethazine 10 mg intravenous administration
  Interventions: Drug: Promethazine
- Saline Placebo (Placebo Comparator): Volume-matched saline placebo
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Ondansetron — 4 mg intravenous dose administered over 2 minutes through a peripheral intravenous catheter
  Arms: Ondansetron
Drug: Metoclopramide — 10 mg intravenous dose administered over 2 minutes through a peripheral intravenous catheter
  Arms: Metoclopramide
Drug: Promethazine — 12.5 mg intravenous dose administered over 2 minutes through a peripheral intravenous catheter
  Arms: Promethazine
Drug: Normal Saline — Volume matched isotonic sodium chloride solution dose administered over 2 minutes through a peripheral intravenous catheter
  Arms: Saline Placebo

SUMMARY:
The purpose of this study is to compare the effectiveness of ondansetron, metoclopramide, and promethazine for the treatment of nausea in the adult emergency department population.

We hypothesize that a single intravenous dose of ondansetron is more effective in reducing nausea than a single IV dose of metoclopramide, promethazine or normal saline placebo in undifferentiated adult emergency department patients.

ELIGIBILITY:
Inclusion Criteria:

* All patients age 18 or older who present to the ED with a complaint requiring antiemetic treatment who do not meet the exclusion criteria.

Exclusion Criteria:

* Patients less than 18 years of age
* Unstable patients with SBP < 90
* Patients with a stated or documented allergy to any of the study medications
* Patients whose nausea rating if < 40 on the pretreatment VAS scale
* Patients who have received a commonly accepted antiemetic within the previous 24 hours
* Patients unwilling or unable to complete the assessment tool before and 30 minutes after study drug dosing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 171 (Actual)
Dates: Start 2007-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tyler W Barrett, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Result] Barrett TW, DiPersio DM, Jenkins CA, Jack M, McCoin NS, Storrow AB, Singleton LM, Lee P, Zhou C, Slovis CM. A randomized, placebo-controlled trial of ondansetron, metoclopramide, and promethazine in adults. Am J Emerg Med. 2011 Mar;29(3):247-55. doi: 10.1016/j.ajem.2009.09.028. Epub 2010 Mar 26. PMID 20825792

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment started March 2007 and completed October 2008. A covenience sample of all adult patients who presented to the emergency department (ED) with a complaint requiring antiemetic treatment who do not meet the exclusion criteria were considered for enrollment.
Pre-assignment Details: Not applicable to this study
Groups:
- Ondansetron: Patients randomized to a single 2 milliliter (mL) Ondansetron 4 mg intravenous dosage administration treatment
- Metoclopramide: Patients randomized to a single 2 mL Metoclopramide 10 mg intravenous dosage administration treatment
- Promethazine: Patients randomized to a single 2 mL Promethazine 12.5mg intravenous dosage administration treatment
- Placebo: Patients randomized to a single 2-mL isotonic sodium chloride Saline Placebo intravenous treatment
Period: Overall Study
Arm/Group | Ondansetron | Metoclopramide | Promethazine | Placebo
Started | 42 | 43 | 45 | 41
Completed | 41 (1 patient withdrawn by treating physician after consent) | 40 (1 patient given drug orally rather than intravenous(iv);1 patient refused iv; 1 pt lost to follow-up) | 43 (1 patient left the ED prior to receiving drug; 1 patient's nausea resolved prior to receiving drug) | 39 (1 patient's initial Visual analog scale (VAS)<40; 1 patient was withdrawn by treating physician)
Not Completed | 1 | 3 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ondansetron | Metoclopramide | Promethazine | Placebo | Total
Number analyzed (Participants) | 42 | 43 | 45 | 41 | 171
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 37 | 40 | 43 | 38 | 158
  >=65 years | 5 | 3 | 2 | 3 | 13
Age Continuous [Mean (Standard Deviation); unit: years] | 39.98 (16.895) | 38.72 (16.076) | 35.47 (16.036) | 35.44 (14.589) | 37.14 (15.882)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 30 | 31 | 27 | 115
  Male | 15 | 13 | 14 | 14 | 56
Region of Enrollment [Number; unit: participants]
  United States | 42 | 43 | 45 | 41 | 171

OUTCOME MEASURES:

1. Primary Outcome: Change in Visual Analog Scale (VAS) Score for Nausea. This Was Calculated by Subtracting the Patient's Reported Score on the 30 Minute VAS From the Patient's Reported VAS Score on Their Baseline VAS.
Description: Participants independently rated their nausea severity on separate scales at the baseline and 30-minute evaluations to prevent the baseline VAS score from influencing the 30-minute mark. The VAS had the words "Least Severe" on the left and "Most Severe" on the right. The possible values range from 0 to 100mm with 0 at the "Least Severe" extreme and 100 at the "Most Severe" extreme. Investigators instructed the participant to draw a single vertical line through the point on the 100mm scale that corresponded to their nausea severity at the times of measurement (Baseline and 30 minutes).
Time Frame: Baseline and 30 minute assessments
Population: Analysis was performed on all patients who received one of the four treatments and completed the 30-minute VAS assessment. The trial was anticipated to require 18 months to achieve full accrual of patients (n=600). Given that we were at 30% information fraction at 17 months, an unplanned interim analysis was done.
Measure: Median (Inter-Quartile Range); unit: millimeter
Arm/Group | Ondansetron | Metoclopramide | Promethazine | Placebo
Number analyzed (Participants) | 41 | 40 | 43 | 39
millimeter | -22.0 [-43.0 to -8.0] | -30.0 [-43.5 to -20.0] | -29.0 [-46.5 to -9.5] | -16.0 [-45.0 to -1.5]
Statistical Analysis 1: Comparison: Ondansetron vs Metoclopramide vs Promethazine vs Placebo; The null hypothesis is that ondanestron is not more effective in reducing nausea than metoclopramide, promethazine or isotonic normal saline. The sample size was chosen to detect a 12-mm difference in VAS improvement between ondanestron and any other treatment arm (assuming a SD of 25mm) at 90% power and 0.01 alpha significance level. We chose the 0.01 alpha level following a Bonferroni type of correction so that the overall type I error rate is about 0.05; Test type: Non-Inferiority or Equivalence — Based on the aforementioned values, we calculated a sample size for each treatment arm of 131 patients. We increased this sample estimate to 150 per treatment arm (total of 600 patients) to account for anticipated study attrition. Based on an unplanned interim conditional power futility analysis done at 30% information fraction, the decision was made to end the trial early.The futility analysis found the observed differences were far less than what was deemed clinically important; p = 0.16, Kruskal-Wallis — Being aware of the multiple comparison issues, we deliberately chose the 0.01 alpha level following a Bonferroni type of correction so that the overall type I error rate is about 0.05; We computed the effect of the 3 treatments relative to ondansetron; Median Difference (Final Values) = 12, Standard Deviation 25 — Change in VAS score was calculated as (VAS 30 min - VAS baseline). We calculated the differences in median VAS reductions for each arm relative to ondansetron

ADVERSE EVENTS:
Arm/Group | Ondansetron | Metoclopramide | Promethazine | Placebo
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/40 | 0/43 | 0/39
Other Adverse Events (participants affected / at risk) | 10/41 | 18/40 | 14/43 | 9/39
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ondansetron (N=41) | Metoclopramide (N=40) | Promethazine (N=43) | Placebo (N=39)
Increased Sedation following treatment (General disorders) | 3 | 12 | 11 | 6 — Patients were asked whether they felt more fatigued or tired.
Pain at iv site following medication administration (Skin and subcutaneous tissue disorders) | 6 | 3 | 6 | 1 — Patients were asked if they experienced burning at the site of their intravenous catheter following drug administration.
Headache following treatment (Nervous system disorders) | 2 | 2 | 1 | 4 — Patients were asked if they experienced a new headache following drug administration?
Akathisia (General disorders) | 0 | 7 | 0 | 0 — Patient was asked if they are feeling abnormally restless or fidgety following drug administration?

LIMITATIONS AND CAVEATS:
Early termination resulted in failure to meet our predetermined sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes